CLINICAL TRIAL: NCT06002529
Title: Hemodiafiltration With Endogenous Reinfusion on Uremic Toxins Clearance of Maintenance Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Renhua Lu, chief physician, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KY2023-077
Record Dates: First submitted 2023-07-10; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: To Evaluate the Clearance Rate of Uremic Toxin by HFR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFR treatment (Other): patient received HFR treatment
  Interventions: Other: HFR

INTERVENTIONS:
Other: HFR — patient received HFR treatment

SUMMARY:
1.1Primary Objective To evaluate the clearance rate of uremic toxin β2-microglobulin (β2-MG), indoxyl sulfate and λ-free light chain (λFLC) by HFR.

1.2Secondary Objectives 1.1.1 To evaluate the clearance of low molecular weight uremic toxin urea (spKt/V, URR).

1.1.2 To evaluate the clearance of other middle molecules and macromolecular uremic toxins, including α1-microglobulin (α1-MG), κ-free light chain (κFLC), homocysteine (Hcy), interleukin-6 (IL-6), p-cresol, YKL-40, complement factor D (CFD), leptin, hippuric acid, trimethylamine oxide (TMAO), asymmetric dimethylarginine (ADMA), tumor necrosis factor-α (TNF- α), myoglobin, fibroblast growth factor 23 (FGF23) and intact parathyroid hormone (iPTH).

1.1.3 To evaluate the clearance of serum albumin, branched chain amino acids and vitamins A, C, E.

1.1.4 To evaluate the comfort of HFR treatment for MHD patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, regardless of gender.
* MHD for at least 3 months, and blood purification treatment for 3 times per week.
* The vascular access is autogenous arteriovenous fistula or artificial blood vessels，with a blood flow ≥200mL/min.
* spKt/V≥1.2.
* Patients who signed the informed consent form (ICF) voluntarily.

Exclusion Criteria:

* Patients who have participated in other interventional clinical trials within a month.
* Pregnant or lactating women.
* Patients of NYHA class IV or occurred acute coronary syndrome or myocardial infarction in 3 months before the start of the study.
* Patients with active hemorrhage in 2 weeks (e.g., cerebral hemorrhage, gastrointestinal hemorrhage, fundus hemorrhage, etc.).
* Patients with unstable blood pressure (pre-dialysis systolic blood pressure ≥180 or ≤90mmHg, pre-dialysis diastolic blood pressure ≥100 or ≤60mmHg), severe anemia (hemoglobin ≤60g/L), and high risk of blood coagulation (e.g., albumin ≤25g/L or hemoglobin ≥140g/L).
* Patients with severe infection (the level of hypersensitive C-reactive protein(hsCRP) ≥ 10×upper limit of normal).
* Patients with a history of drug addiction or severe mental disorders.
* Other conditions in which the investigators reject patients to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-18 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
β2-microglobulin (β2-MG), indoxyl sulfate and λ-free light chain (λFLC) | 1 day
  The concentrations of β2-microglobulin (β2-MG), indoxyl sulfate and λ-free light chain (λFLC) were measured before and after HFR

SECONDARY OUTCOMES:
Single-compartment urea clearance index (spKt/V), Urea Reduction Ratio | 1 day
  Calculate spKt/V and Urea Reduction Ratio.
other middle molecules and macromolecular uremic including α1-MG, κFLC, Hcy, IL-6, p-cresol, YKL-40, CFD, leptin, hippuric acid, TMAO, ADMA, TNF-α, myoglobin, FGF23 and iPTH | 1 day
  The concentrations of other middle molecules and macromolecular uremic were measured before and after HFR
serum albumin, branched chain amino acids and vitamins A, C, E | 1 day
  The concentrations of serum albumin, branched chain amino acids and vitamins A, C, E before and after HFR
the comfort of HFR treatment | 1 day
  The dialysis comfort score was used for evaluation

IPD SHARING:
Plan to Share IPD: No